CLINICAL TRIAL: NCT04384393
Title: A Study to Evaluate the Safety and Clinical Activity of Allogeneic Chimeric Antigen Receptor T Cells Targeting CD19 in Patients With Refractory or Relapsed B Cell Malignancies.
Brief Title: Safety and Efficacy of ThisCART19 in Patients With Refractory or Relapsed B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundamenta Therapeutics, Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART19
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: B Cell Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19 cells injections (Experimental): In this study, allogeneic anti-CD19 CAR T Cells(ThisCART19 cells) is used to treat patients with refractory or relapsed CD19 positive B cell malignancies.
  Interventions: Biological: ThisCART19 cells

INTERVENTIONS:
Biological: ThisCART19 cells — 0.2-60 x 10^6 CAR T cells per kg body weight.

SUMMARY:
This is a study to evaluate the safety and clinical activity of ThisCART19 (Allogeneic CAR-T targeting CD19) in patients with refractory or relapsed CD19 positive B cell malignancies.

DETAILED DESCRIPTION:
This is a single-center, nonrandomized, open-label study to evaluate the safety and clinical activity of ThisCART19 in patients with refractory or relapsed CD19 positive B cell malignancies, such as acute or chronic lymphocytic leukemia, lymphoma and etc. The dose range is 0.2-60 x 10^6 cells per kg body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with relapsed or refractory CD19 positive acute or chronic lymphocytic leukemia, or lymphoma.
2. No alternative treatment options deemed by investigator.
3. Measurable or detectble disease at time of enrollment.
4. Eastern cooperative oncology group (ECOG) performance status of ≤2.
5. Cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO).
6. Estimated life expectancy > 12 weeks deemed by investigator.
7. Serum creatinine ≤1.6 mg/dl and/or blood urea nitrogen(BUN) ≤ 1.5 mg/dl .
8. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 upper limit of normal (ULN).
9. Informed consent explained to, understood by and signed by patient/guardian.

Exclusion Criteria:

1. Pregnant or lactating women
2. Uncontrolled infection
3. Active hepatitis B virus or hepatitis C virus infection.
4. Patients who need steroids to control disease.
5. Patients who accepted autologous stem-cell transplantation (ASCT) within 100 days.
6. Patients with grade 2-4 graft-versus-host disease (GVHD), or deemed need to manage by investigator.
7. History of Human Immunodeficiency Virus (HIV) infection.
8. Patients with active central nervous system (CNS) involvement by malignancy.
9. Patients combine with other disease cause neutrophil count (ANC) < 750 per microlitre or platelet count (PLT)< 50,000 per microlitre.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2023-10-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | From infusion to Day 28
  To assess adverse events as dose limiting toxicities as defined by the protocol.
Complete Remission | At Day 28 after ThisCART19 infusion
  Proportion of patients in whom with morphologic complete remission (CR)
TRM: Treatment Related Mortality | Up to 2 years
  The mortality related with ThisCART19 infusion.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 1 year
  For Acute Lymphoblastic Leukemia (ALL), Objective response rate(ORR) is the percentage of patients who achieve CR or chronic lymphocytic leukemia(CRi); for chronic lymphocytic leukemia (CLL) and lymphoma, ORR is the incidence of either a complete response (CR) or a partial response (PR).
Duration of Response | Up to 1 year
  Duration of Response (DOR) defined as the duration (days) from initial response to disease relapse, progression, or death due to any course.
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | From inclusion up to 1 year
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Overall Survival Rate of 2 Years | At year 2
  The rate of patients whom alive at year 2

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (2):
- China (2):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Fundamenta Therapeutice Co.,Ltd, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No